CLINICAL TRIAL: NCT01870882
Title: Attention Training for Opioid-maintained Cocaine Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1303011711
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Addiction; Cocaine; Methadone; Opiates
Keywords: Opioid-Related Disorders; Cocaine-Related Disorders; Substance-Related Disorders; Mental Disorders; Cocaine; Methadone; Therapeutic Uses
MeSH Terms: conditions — Behavior, Addictive; Opioid-Related Disorders; Cocaine-Related Disorders; Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retraining (Active Comparator): Using the PED, participants repeatedly complete a version of attentional bias task that orients their attention away from drug-related cues.
  Interventions: Behavioral: Attentional retraining
- Control (Sham Comparator): Using the PED, participants repeatedly complete versions of the attentional bias task in which their attention is oriented toward and away from drug-related cues on an equal number of trials.
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: Attentional retraining
  Other Names: attentional training; attentional bias retraining
  Arms: Retraining
Behavioral: Control condition
  Arms: Control

SUMMARY:
The purpose of this study is to determine the feasibility and preliminary efficacy of attention training using a portable electronic device for opioid-dependent cocaine-users stabilized on methadone.

DETAILED DESCRIPTION:
The investigators propose to test the feasibility and preliminary efficacy of 5-times per week daily attentional retraining (AR) delivered via a portable electronic device (PED) in comparison with a control condition over the course of a 2-3 week training period. Participants in this study will be cocaine and opioid-dependent individuals stabilized on methadone. Both cocaine and opioids will be targeted in the AR procedure the investigators will test in this study. The retraining or control condition, along with a series of assessments, will be delivered on the PED as part of a daily (Monday through Friday) appointment at which time participants will also obtain their daily methadone dose. Assessments will cover substance use, craving and other issues. In addition to completing the retraining or control procedure, participants will also be engaged in standard versions of attentional bias tasks (i.e., without retraining) periodically in order to gauge an effect of study condition on attentional bias over time. Thus, the investigators will be able to track changes in attentional bias over time in a more detailed fashion than has been previously possible. Following the 3 week training period, there will be another 3 weeks of treatment in which patients will continue to receive methadone and complete limited assessments without any AR or control procedures with the PED.

ELIGIBILITY:
Inclusion Criteria:

* Current opioid dependence as evidenced by 1) documentation of prior treatment for opioid dependence or signs of withdrawal, 2) self-reported history of opioid dependence for 12 consecutive months and, 3) a positive urine toxicology screen for opiates.
* Diagnosis of opioid dependence and cocaine dependence as well as laboratory confirmation of recent cocaine use in the form of positive urine toxicology during the month prior to study entry.
* For those who recently participated in a research study involving medications other than methadone, at least 2 weeks of washout period before enrollment. Those already taking methadone would continue with their current course while participating in this study.
* A history of cocaine use, a minimum of 1/2 gram and more than once per week during the preceding 30 days.
* Must be seeking treatment for opioid and cocaine use.
* For women of childbearing age, a negative pregnancy test at screening with agreement to use adequate contraception to prevent pregnancy and monthly pregnancy tests.
* The ability to speak, read, and write in English at an eight-grade literacy level.

Exclusion Criteria:

* Serious medical illnesses including hypertension, tachycardia, bradycardia, or other arrhythmias and major cardiovascular, cerebrovascular, renal, endocrine, or hepatic disorders;
* Serious psychiatric illness, history of psychosis, schizophrenia or bipolar type I disorder.
* Current major depression. Subjects with current depressive symptoms not meeting criteria will be included in the study, with the exception of those endorsing suicidal and homicidal thoughts, will be excluded even if full criteria for major depression are not met.
* Current diagnosis of alcohol or drug dependence other than opiates, cocaine, nicotine and cannabis.
* Current use of over-the-counter or prescription psychoactive drugs (antidepressant, anxiolytics, antipsychotics, mood stabilizers, psychostimulants) or drugs that would be expected to have major interactions with drugs to be tested, e.g., benzodiazepines, codeine, percocet, and other opiate drugs that will interact with methadone.
* Liver function tests (ALT or AST) greater than 3 times normal.
* Self-reported color blindness or (non-corrected) defective vision

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Attentional bias for cocaine cues | over the course of the 3 week training period
  The tendency to respond more rapidly to a dot probe when the probe replaces a cocaine-related word than when a dot probe replaces a matched, non-drug control word.
Attentional bias for opioid cues | over the course of the 3 week training period
  The tendency to respond more rapidly to a dot probe when the probe replaces an opioid-related word than when a dot probe replaces a matched, non-drug control word.
Retention of participants in treatment | at the end of the 3 week training period
Mean duration of sessions with the PED | the duration of the 3 week training period

SECONDARY OUTCOMES:
self-reported craving for cocaine | assessed on a daily basis during the 3 week training period
Self-reported cocaine use | during the 3 week training period
Self-reported opioid use | during the 3 week training period
self-reported craving for opiates | assessed on a daily basis during the 3 week training period
Cocaine urine test results | during the 3 week training period
opioid urine test results | during the 3 week training period

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Leeman, Ph.D., Principal Investigator — Yale University
Locations (1):
- Department of Veterans Affairs Hospital, West Haven, Connecticut, United States